CLINICAL TRIAL: NCT02397018
Title: Allogeneic Umbilical Cord Blood Infusion for Adults With Ischemic Stroke
Brief Title: Cord Blood Infusion for Ischemic Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joanne Kurtzberg, MD (Other)
Responsible Party: Sponsor-Investigator, Joanne Kurtzberg, MD, Principal Investigator, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00059284
Record Dates: First submitted 2015-03-19; First posted 2015-03-24 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Stroke
Keywords: stroke; cord blood; umbilical cord blood; hematopoietic stem cells; acute ischemic stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic Umbilical Cord Blood Infusion (Experimental): All subjects in this study will receive an intravenous infusion of ABO/Rh matched umbilical cord blood.
  Interventions: Biological: allogeneic umbilical cord blood

INTERVENTIONS:
Biological: allogeneic umbilical cord blood — Umbilical cord blood units will be selected from a public cord blood bank based on ABO/Rh blood type and cell dose, targeting a range of 0.5 to 5 x 10^7 total nucleated cells per kilogram. The cord blood unit will be intravenously infused into the subject over 5-30 minutes at a rate not exceeding 5 mL/kg/hr. Subjects will not receive immunosuppressive medications or any other cytoreduction prior to infusion.
  Other Names: cord blood; umbilical cord blood

SUMMARY:
This is a phase one study investigating the safety of a single, intravenous infusion of banked allogeneic umbilical cord blood in subjects following an acute ischemic stroke. The cord blood infusion must be given within 3-10 days of the stroke. Follow up phone calls will occur at 1, 6, and 12 months post-infusion, and will include telephone surveys on post-stroke rehabilitation and functioning. A follow up clinic visit at 90 days will include a neurological exam, MRI, and blood tests.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety of a single, intravenous infusion of banked allogeneic umbilical cord blood in subjects within 3-10 days following an acute ischemic stroke. The subjects will not be pre-treated with immunosuppressive agents. The primary objective is safety assessment and the secondary objectives are to determine which outcome measures can be used as primary and secondary endpoints for future randomized Phase 2 clinical trials, and to describe clinical responses, if any. All subjects will receive standard of care acute and rehabilitation treatments while enrolled in this study.

This is a multicenter Phase 1 safety study in patients 18-80 years of age who have sustained a recent ischemic stroke. A total of 10 subjects will be enrolled. Subjects will be given a series of baseline neurological assessments, blood tests, and MRI. Umbilical cord blood units will be selected from a public cord blood bank based on ABO/Rh blood type and cell dose, targeting a range of 0.5 to 5 x 10^7 total nucleated cells/kg. Umbilical cord blood will be administered intravenously as a single infusion between 3 and 10 days post-stroke. Subjects will be monitored for 6 hours post-infusion, and follow up will occur 24 hours later. Subsequent follow up phone calls will occur at 1, 6, and 12 months, and will include telephone surveys on post-stroke rehabilitation and functioning. A follow up clinic visit at 90 days will include a neurological exam, MRI, and blood tests.

Risks of cord blood infusion include infusion-related reactions such as anaphylaxis, urticaria, dyspnea, hypoxia, cough, wheezing, bronchospasm, nausea, vomiting, hives, fever, hypertension, hypotension, bradycardia, tachycardia, rigors, chills, infection, and hemoglobinuria. Less likely, long-term risks include transmission of infection or Graft vs Host Disease.

ELIGIBILITY:
Inclusion Criteria:

An individual is eligible for inclusion if all of the following apply:

1. Is 18-80 years old
2. Has had a recent (within the past 9 days), acute, cortical, hemispheric, ischemic stroke in the middle cerebral artery (MCA) distribution without a midline shift as detected by magnetic resonance imaging (MRI) as a diffusion-weighted image (DWI) abnormality
3. Has a National Institutes of Health Stroke Scale (NIHSS) score of 8-15 (R) and 8-18 (L) at the time of enrollment with no more than a 4 point increase (worsening of score) from the baseline score compared to 24 hours prior to infusion
4. Subjects must have a platelet count >100,000/uL, hemoglobin >8gm/dl, and white blood cell count (wbc) >2,500/uL.
5. Subjects who received tissue plasminogen activator (tPA) or underwent mechanical reperfusion may be included in the study.
6. Is able to provide consent to study or consent is obtained from the subject's legally authorized representative
7. Subjects of childbearing potential must practice effective contraception during the study, and be willing to continue contraception for at least 6 months after intervention so that, in the opinion of the investigator, they will not become pregnant during the course of the study
8. Is a good candidate for the trial, in the opinion of the investigator
9. Agrees to participate in follow up visits
10. Has an ABO/Rh matched umbilical cord blood unit with a minimum of 0.5 x 10^7 total nucleated cells (TNCC)/kg based on the pre-cryopreservation TNCC.

Exclusion Criteria:

An individual is ineligible to participate if any of the following apply.

Medical Conditions:

1. Has a medical history of neurological or orthopedic pathology with a deficit as a consequence that results in a modified Rankin Scale >1 before stroke or has a pre-existing cognitive deficit
2. Has clinically significant and/or symptomatic hemorrhage associated with stroke
3. Has new intracranial hemorrhage, edema, or mass effect that may place patient at increased risk for secondary deterioration when assessed prior to infusion
4. Has hypotension as defined as the need for IV pressor support of systolic blood pressure <90
5. Has isolated brain stem stroke
6. Has pure lacunar stroke
7. Requires mechanical ventilation
8. Requires a craniotomy
9. Has a serious psychiatric or neurological disease which could alter evaluation on functional or cognitive scales
10. Has an active systemic infection or is HIV positive
11. Has had an active malignancy within 3 years prior to the start of screening excluding skin cancers other than melanoma
12. Has known coagulopathy such as Factor V Leyden, AntiPhospholipid Syndrome (APC), Protein C, Protein S deficiency, sickle cell, anticardiolipin antibody, or phospholipid syndrome
13. Has any concurrent illness or condition that in the opinion of the investigator might interfere with treatment or evaluation of safety
14. Has current or recent history of alcohol or drug abuse, or stroke associated with drug abuse
15. Pregnant as documented by urine or blood test

Concomitant or Prior Therapies:

1. Subjects currently receiving immunosuppressant drugs
2. History of prior transfusion reaction
3. Currently on dialysis
4. Recipient of bone marrow or organ transplant
5. Renal insufficiency with serum creatinine >2.0 mg/dL
6. Hepatic insufficiency (bilirubin >2.5mg/dL or transaminases >5x the upper limit of normal). Patients with Gilberts syndrome are eligible for study enrollment if other liver function tests are normal, regardless of bilirubin level.
7. Any previous or current treatment with angiogenic growth factors, cytokines, gene or stem cell therapy
8. Subjects participating in another interventional clinical trial of an investigational therapy within 30 days of screening

Other:

1. Pregnant or lactating women
2. Unable to be evaluated for follow up visits

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05; Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 12 months post-infusion for the last subject
  Number of subjects experiencing any study related Adverse Event (AE) during the 12-month follow-up period
Graft Versus Host Disease | 100 days
  The proportion of subjects experiencing Graft Versus Host Disease (GVHD) at Day 100 post-infusion

SECONDARY OUTCOMES:
Change in modified Rankin Score | 3 months post-infusion for the last subject
  The mean change in modified Rankin Score from baseline to 3 months post-infusion
Change in Infarct Volumes | 3 months post-infusion for the last subject
  Describe changes in infarct volumes over the first 3 months post-stroke

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Kurtzberg, M.D., Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Houston Methodist, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Laskowitz DT, Bennett ER, Durham RJ, Volpi JJ, Wiese JR, Frankel M, Shpall E, Wilson JM, Troy J, Kurtzberg J. Allogeneic Umbilical Cord Blood Infusion for Adults with Ischemic Stroke: Clinical Outcomes from a Phase I Safety Study. Stem Cells Transl Med. 2018 Jul;7(7):521-529. doi: 10.1002/sctm.18-0008. Epub 2018 May 12. PMID 29752869